CLINICAL TRIAL: NCT06368518
Title: Austrian Hypertrophic Cardiomyopathy Registry
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Nicolas Dominik Verheyen, MD, Principal Investigator, Medical University of Graz
Other Study IDs: ID01/2024/MZHCM-Reg/NV
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic Cardiomyopathy; Left ventricular hypertrophy; Hypertrophic Phenotype
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Austrian Hypertrophic Cardiomyopathy (HCM) Registry is a prospective, multicenter registry enrolling patients at multiple outpatient clinics across Austria including academic and non-academic centers. Patients will undergo a structured examination process including assessment for symptoms of HCM, past medical history, concomitant medication, family history and the presence of HCM-specific red flags. Furthermore, clinical data derived from electrocardiogram, echocardiography, laboratory analysis, and genetic testing will be collected focusing on a lean variable dictionary and, in addition, specific hypothesis-driven research parameters. All data are entered into an electronic case report form (eCRF) (Phoenix Clinical Trial Management System). In order to perform multicenter analyses, data can be extracted from the eCRF after approval by the steering committee.

DETAILED DESCRIPTION:
The Austrian Hypertrophic Cardiomyopathy (HCM) Registry is a prospective, multicenter registry enrolling patients at multiple outpatient clinics across Austria including academic and non-academic centers. Patients will undergo a structured examination process including assessment for symptoms of HCM, past medical history, concomitant medication, family history and the presence of HCM-specific red flags. Furthermore, clinical data derived from electrocardiogram, echocardiography, laboratory analysis, and genetic testing will be collected focusing on a lean variable dictionary and, in addition, specific hypothesis-driven research parameters. All data are entered into an electronic case report form (eCRF) (Phoenix Clinical Trial Management System). Every site will nominate one representative for the steering committee which will serve as the regulatory authority with the compentence to approve research and funding proposals.

The Austrian multicenter HCM Registry aims to facilitate a wide range of innovative cross-sectional and longitudinal epidemiological analyses unravelling gaps in evidence in HCM. The standardized clinical assessment might harmonize standards of clinical care in HCM patients in Austria.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the HCM outpatient clinic of participating centers of the HCM Registry
* Interventricular septal thickness ≥ 13 mm and cardiomyopathy-specific red flags OR Interventricular septal thickness ≥ 15 mm not explainable by loading conditions OR Interventricular septal thickness ≥ 17 mm
* Willingness and ability to provide signed informed consent form (ICF) prior to participation in any study-related procedures

Exclusion criteria:

* Age < 18 years
* Known cardiac amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects who fulfill criteria of HCM and are treated in Austria.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2044-03 (Estimated); Study Completion 2044-03 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Through study completion, on average 20 years
  All cause mortality
Cardiovascular events | Through study completion, on average 20 years
  Cardiovascular events

CONTACTS AND LOCATIONS:
Locations (15):
- Austria (15):
  - Kepler University Hospital Linz, Linz, Linz
  - University Hospital St. Pölten, Sankt Pölten, Lower Austria
  - Hospital Landesklinikum Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Paracelsus Medical University of Salzburg, Salzburg, Salzburg
  - Clinic Cardinal Schwarzenberg, Schwarzach im Pongau, Salzburg
  - Hospital Graz 2 West, Graz, Styria
  - Medical University of Graz, Graz, Styria
  - Medical University of Innsbruck, Innsbruck, Tyrol
  - Hospital St. Josef Braunau, Braunau am Inn, Upper Austria
  - Ordensklinikum Linz, Linz, Upper Austria
  - Medical University of Vienna, Vienna, Vienna
  - Favoriten Clinic Vienna, Vienna, Vienna
  - Klinik Ottakring, Vienna, Vienna
  - General Hospital St. Johann in Tirol, Sankt Johann in Tirol
  - Clinic Wels-Grieskirchen, Wels-Grieskirchen